CLINICAL TRIAL: NCT01140958
Title: A Retrospective Pharmacoeconomic Study of Lung Cancer in Wan-Fang Hospital
Brief Title: A Retrospective Pharmacoeconomic Study of Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hsingjin Eugene Liu, MD PhD, Taipei Medical University WanFang Hospital
Other Study IDs: Pharmacoeconomic-01
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Lung Cancer
Keywords: lung cancer; pharmacoeconomics; new agents
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Lung cancer is the No. cause of cancer death in Taiwan. Yet most of lung cancer are diagnosed at late stage, not amenable to surgical resection. With the introduction of new targeted agents, such as EGFR tyrosine kinase inhibitors and the identification of EGFR mutations, lung cancer management has markedly changed in recent years. However, these new agents are costly and their payment is restricted in certain situations defined National Insurance Agency. Therefore, using databases from National Insurance Agency might not be able to reflect the exact impact on pharmacoeconomics. In this study, the investigators will analyze the data from a tertiary medical center, where all the costs including insurance reimbursement, co-payment, and payment not covered by insurance. The investigators will also compare with the investigators results with national database to analyze the cost benefit of these new agents on lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer patients in WanFang Hospital

Exclusion Criteria:

* non

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: lung cancer patients in WanFang Hospital
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Gjin Eugene Liu, Principal Investigator — Taipei Medical University WanFang Hospital